CLINICAL TRIAL: NCT02986178
Title: A Multicenter Phase 2 Study of Oncolytic Polio/Rhinovirus Recombinant (Lerapolturev) in Recurrent WHO Grade IV Malignant Glioma Patients
Brief Title: Lerapolturev in Recurrent Malignant Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Istari Oncology, Inc. (Industry)
Collaborators: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00077024
Record Dates: First submitted 2016-12-06; First posted 2016-12-08 (Estimated); Results first posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-04

CONDITIONS: Malignant Glioma
Keywords: Glioblastoma; Glioma; PVSRIPO; Duke; Pro00077024; Brain tumor; Istari; Recurrent; GBM; rGBM
MeSH Terms: conditions — Glioma; Glioblastoma; Brain Neoplasms; Recurrence | interventions — Lomustine

STUDY DESIGN:
Intervention Model Description: Study began as parallel (randomized two arm study) and was revised to single group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- lerapolturev (Experimental): lerapolturev administered once intratumorally by convection-enhanced delivery
  Interventions: Biological: lerapolturev
- lerapolturev + lomustine (Experimental): lerapolturev administered once intratumorally by convection-enhanced delivery plus one dose of lomustine at 8 weeks post-lerapolturev dosing
  Interventions: Biological: lerapolturev; Drug: Lomustine

INTERVENTIONS:
Biological: lerapolturev — A single dose of lerapolturev, an oncolytic polio/rhinovirus recombinant
  Other Names: PVSRIPO
Drug: Lomustine — one cycle of oral lomustine
  Other Names: gleostine
  Arms: lerapolturev + lomustine

SUMMARY:
This is a phase 2 study of lerapolturev, an oncolytic polio/rhinovirus recombinant, in adult patients with recurrent World Health Organization (WHO) grade IV malignant glioma.

DETAILED DESCRIPTION:
This is a Phase 2 study of lerapolturev, an oncolytic polio/rhinovirus recombinant, in adult patients with recurrent World Health Organization (WHO) grade IV malignant glioma. The objective of this study is to investigate the safety and efficacy (anti-tumor response and survival) of lerapolturev in recurrent WHO grade IV malignant glioma.

Patients will be administered lerapolturev intratumorally via convection-enhanced delivery (CED) using an intracerebral catheter placed within the enhancing portion of the tumor. Retreatment with lerapolturev is allowed, provided retreatment eligibility criteria are met.

ELIGIBILITY:
INCLUSION CRITERIA SUMMARY:

1. Patients must have a recurrent (first or second recurrence only, including this recurrence; transformation from a lower grade tumor to a WHO grade IV malignant glioma will be considered a first recurrence) supratentorial WHO grade IV malignant glioma based on imaging studies with measurable disease (a minimum measurement of 1 cm and maximum of 5.5 cm of contrast-enhancing tumor) with prior histopathology consistent with a WHO grade IV malignant glioma confirmed by the site's neuropathologist or the neuropathologist's designate.
2. Male patients who are sexually active are eligible if he and/or his partner(s) meets the criteria outlined in the protocol. Female subjects are eligible if he and/or his partner(s) meets the criteria outlined in the protocol.
3. Age ≥ 18 years of age.
4. Karnofsky Performance Status (KPS) Score ≥ 70%.
5. Prothrombin and Partial Thromboplastin Times ≤ 1.2 x normal prior to biopsy.
6. Total bilirubin, serum glutamic oxaloacetic transaminase (SGOT), serum glutamic pyruvic transaminase (SGPT), alkaline phosphatase ≤ 2.5 x normal prior to biopsy.
7. Neutrophil count ≥ 1000 prior to biopsy.
8. Hemoglobin ≥ 9 prior to biopsy.
9. Platelet count ≥ 100,000/μL unsupported is necessary for eligibility on study; however, because of risks of intracranial hemorrhage with catheter placement, platelet count ≥ 125,000/μL is required for the patient to undergo biopsy and catheter insertion, which can be attained with the help of platelet transfusion.
10. Creatinine ≤ 1.2 x normal range prior to biopsy.
11. Positive serum anti-PV titer prior to biopsy.
12. The patient must have received a boost immunization with trivalent inactivated IPOL™ (Sanofi-Pasteur) at least 1 week, but less than 6 weeks, prior to administration of the study agent.
13. At the time of biopsy, prior to administration of virus, the presence of recurrent tumor must be confirmed by histopathological analysis.
14. A signed IRB-approve informed consent form (ICF).
15. Able to undergo brain MRI with and without contrast.

EXCLUSION CRITERIA SUMMARY:

1. Females who are pregnant or breast-feeding.
2. Patients with an impending, life-threatening cerebral herniation syndrome, based on the assessment of the study neurosurgeons, their designate, and the reviewer designated by the sponsor.
3. Patients with severe, active co-morbidity, defined as in the protocol.
4. Patients with a previous history of neurological complications due to PV infection.
5. Patients who have not recovered from the toxic effects of prior chemo- and/or radiation therapy. Guidelines for this recovery period are dependent upon the specific therapeutic agent being used.
6. Patients may not have received tumor treating fields (≤ 1 week), chemotherapy or bevacizumab ≤ 4 weeks [except for nitrosourea and lomustine (≤ 6 weeks); metronomic dosed chemotherapy, such as daily temozolomide, etoposide or cyclophosphamide (≤ 1 week)] prior to starting the study drug.
7. Patients may not have received immunotherapy ≤ 4 weeks prior to starting the study drug unless patients have recovered from side effects of such therapy.
8. Patients may not be less than 12 weeks from radiation therapy of the brain, unless progressive disease outside of the radiation field or 2 progressive scans at least 4 weeks apart or histopathologic confirmation.
9. Prior to enrollment, has not completed all standard of care treatments, including surgical procedure and radiation therapy (at least 59Gy) as outlined in the protocol.
10. Patients with neoplastic lesions in the brainstem, cerebellum, or spinal cord; radiological evidence of multiple areas of active (growing) disease (active multifocal disease); tumors with contrast-enhancing tumor component crossing the midline (crossing the corpus callosum); extensive subependymal disease (tumor touching subependymal space is allowed); or extensive leptomeningeal disease (tumor touching leptomeninges is allowed).
11. Patients with undetectable anti-tetanus toxoid immunoglobulin G (IgG).
12. Patients with known history of agammaglobulinemia.
13. Patients on greater than 4 mg per day of dexamethasone within the 2 weeks prior to admission for lerapolturev infusion.
14. Patients with worsening steroid myopathy (history of gradual progression of bilateral proximal muscle weakness, and atrophy of proximal muscle groups).
15. Patients with prior, unrelated malignancy requiring current active treatment with the exception of cervical carcinoma in situ and adequately treated basal cell or squamous cell carcinoma of the skin.
16. For patients randomized prior to V7, a known history of hypersensitivity to lomustine, dacarbazine, or any components of lomustine.
17. Patients with active autoimmune disease requiring systemic immunomodulatory treatment within the past 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-02-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Head of Clinical Operations, Study Director — Istari Oncology
Locations (6):
- United States (6):
  - UCSF Neurological Surgery, San Francisco, California
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Preston Robert Tisch Brain Tumor Center at Duke University, Durham, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brown MC, Beasley GM, McKay ZP, Yang Y, Desjardins A, Randazzo DM, Landi D, Ashley DM, Bigner DD, Nair SK, Gromeier M. Intratumor childhood vaccine-specific CD4+ T-cell recall coordinates antitumor CD8+ T cells and eosinophils. J Immunother Cancer. 2023 Apr;11(4):e006463. doi: 10.1136/jitc-2022-006463. PMID 37072349
- See also: The Preston Robert Tisch Brain Tumor Center at Duke University — https://tischbraintumorcenter.duke.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The lerapolturev + lomustine arm was closed after interim review. Recruitment to the lerapolturev alone arm remained open.
Pre-assignment Details: Safety set includes all enrolled participants who had an infusion catheter placed.
  Full-analysis set includes all randomized participants who received lerapolturev treatment.
Groups:
- Not Treated: Includes a participant who had an infusion catheter placed but withdrew from the study prior to receiving lerapolturev.
Period: Overall Study
Arm/Group | Lerapolturev | Lerapolturev + Lomustine | Not Treated
Started | 93 | 27 | 1
Completed | 93 | 27 | 0
Not Completed | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Data are reported on the Full Analysis Set which includes participants that were randomized, had an infusion catheter placed, and received the initial dose of lerapolturev. The full analysis set is 120 participants. Data are not reported on the single participant who was consented, had an infusion catheter placed and did not receive lerapolturev.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lerapolturev | Lerapolturev + Lomustine | Total
Number analyzed (Participants) | 93 | 27 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (12.4) | 50 (13.6) | 54 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 11 | 39
  Male | 65 | 16 | 81
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 87 | 27 | 114
  Unknown or Not Reported | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 1 | 5
  White | 83 | 26 | 109
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 0 | 5
Region of Enrollment [Number; unit: participants]
  United States | 93 | 27 | 120
Karnofsky Performance Status [Count of Participants; unit: Participants] — The Karnofsky Performance Status is a scale used to measure a patient's ability to perform daily activities. Scores range from 0 to 100 with higher scores indicating better ability to perform daily activities.
  Participants
    70 | 5 | 0 | 5
    80 | 21 | 8 | 29
    90 | 60 | 17 | 77
    100 | 7 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Objective Radiographic Response
Description: Assess objective anti-tumor response based on iRANO criteria.
Time Frame: up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Lerapolturev | Lerapolturev + Lomustine
Number analyzed (Participants) | 93 | 27
Participants | 5 | 2

2. Primary Outcome: Duration of Objective Radiographic Response
Description: Assess time of confirmed response to confirmed disease progression or death
Time Frame: up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lerapolturev | Lerapolturev + Lomustine
Number analyzed (Participants) | 5 | 2
months | NA [NA to NA] — NA = None of the participants with a confirmed response had documented disease progression or death; therefore, the DOR estimates were deemed not estimable (NE). The value "NA" has been entered as the system requires a numerical entry (ie, NE for not estimable cannot be entered). | NA [NA to NA] — NA = None of the participants with a confirmed response had documented disease progression or death; therefore, the DOR estimates were deemed not estimable (NE). The value "NA" has been entered as the system requires a numerical entry (ie, NE for not estimable cannot be entered).

3. Secondary Outcome: Median Overall Survival
Description: Overall Survival (months), calculated using the Kaplan-Meier method
Time Frame: up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lerapolturev | Lerapolturev + Lomustine
Number analyzed (Participants) | 93 | 27
months | 7.0 [5.8 to 9.1] | 7.1 [4.0 to 8.1]

4. Secondary Outcome: Landmark Survival
Description: Overall survival (months) at 24 and 36 months, calculated using the Kaplan-Meier method
Time Frame: at 24 and 36 months post-lerapolturev infusion
Measure: Number (95% Confidence Interval); unit: proportion probability
Arm/Group | Lerapolturev | Lerapolturev + Lomustine
Number analyzed (Participants) | 93 | 27
proportion probability
  Probability of being alive at 24 months | 0.12 [0.06 to 0.21] | 0.19 [0.07 to 0.35]
  Probability of being alive at 36 months | 0.07 [0.02 to 0.15] | 0.11 [0.03 to 0.26]

5. Secondary Outcome: Disease Control Rate
Description: the percentage of participants achieving complete response, partial response, or stable disease
Time Frame: up to 5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lerapolturev | Lerapolturev + Lomustine
Number analyzed (Participants) | 93 | 27
percentage of participants | 51 [40 to 61] | 48 [29 to 68]

6. Secondary Outcome: Safety of Lerapolturev
Description: Number of participants experiencing Grade 3, 4 or 5 adverse events considered possibly, probably, or definitely related to protocol treatment
Time Frame: up to 52 weeks
Population: The safety set includes all participants who had an infusion catheter placed.
Measure: Count of Participants; unit: Participants
Arm/Group | Lerapolturev | Lerapolturev + Lomustine
Number analyzed (Participants) | 94 | 26
Participants | 17 | 8

ADVERSE EVENTS:
Time Frame: Adverse events were collected until study discontinuation, up to 5 years.
Description: The safety set includes all enrolled participants who had an infusion catheter placed. Participants are displayed based on actual treatment received.
Groups:
- Overall: includes a participant who had an infusion catheter placed and did not receive lerapolturev
Arm/Group | Lerapolturev | Lerapolturev + Lomustine | Overall
All-Cause Mortality (participants affected / at risk) | 8/94 | 4/26 | 12/121
Serious Adverse Events (participants affected / at risk) | 37/94 | 12/26 | 50/121
Other Adverse Events (participants affected / at risk) | 94/94 | 26/26 | 121/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lerapolturev (N=94) | Lerapolturev + Lomustine (N=26) | Overall (N=121)
hemiparesis (Nervous system disorders) | 8 | 6 | 14
seizure (Nervous system disorders) | 9 | 5 | 14
aphasia (Nervous system disorders) | 6 | 0 | 6
haemorrhage intracranial (Nervous system disorders) | 6 | 0 | 6
brain oedema (Nervous system disorders) | 2 | 1 | 4
hydrocephalus (Nervous system disorders) | 2 | 0 | 2
ataxia (Nervous system disorders) | 1 | 0 | 1
encephalopathy (Nervous system disorders) | 1 | 0 | 1
somnolence (Nervous system disorders) | 0 | 1 | 1
sepsis (Infections and infestations) | 4 | 1 | 5
urinary tract infection (Infections and infestations) | 5 | 0 | 5
abdominal abscess (Infections and infestations) | 0 | 1 | 1
anorectal infection (Infections and infestations) | 0 | 1 | 1
Ludwig angina (Infections and infestations) | 0 | 1 | 1
respiratory tract infection (Infections and infestations) | 0 | 1 | 1
skin infection (Infections and infestations) | 1 | 0 | 1
embolism (Vascular disorders) | 5 | 3 | 8
haematoma (Vascular disorders) | 1 | 0 | 1
confusional state (Psychiatric disorders) | 4 | 2 | 6
depression (Psychiatric disorders) | 1 | 0 | 1
fatigue (General disorders) | 3 | 0 | 3
cyst (General disorders) | 1 | 0 | 1
localised edema (General disorders) | 1 | 0 | 1
pain (General disorders) | 1 | 0 | 1
pyrexia (General disorders) | 1 | 0 | 1
peritumoral oedema (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 2
gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
gastric haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 1
haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
large intestine perforation (Gastrointestinal disorders) | 1 | 0 | 1
lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
cardiac arrest (Cardiac disorders) | 3 | 0 | 3
fall (Injury, poisoning and procedural complications) | 2 | 0 | 2
rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1
muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
urinary incontinence (Renal and urinary disorders) | 1 | 1 | 2
aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
platelet count decreased (Investigations) | 0 | 1 | 1
headache (Nervous system disorders) | 3 | 5 | 8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lerapolturev (N=94) | Lerapolturev + Lomustine (N=26) | Overall (N=121)
headache (Nervous system disorders) | 63 | 22 | 85
hemiparesis (Nervous system disorders) | 63 | 22 | 85
seizure (Nervous system disorders) | 40 | 17 | 57
aphasia (Nervous system disorders) | 35 | 9 | 44
memory impairment (Nervous system disorders) | 22 | 4 | 26
cognitive disorder (Nervous system disorders) | 15 | 3 | 18
paraesthesia (Nervous system disorders) | 11 | 5 | 16
dizziness (Nervous system disorders) | 9 | 6 | 15
tremor (Nervous system disorders) | 9 | 1 | 10
hemianopia (Nervous system disorders) | 7 | 2 | 9
haemorrhage intracranial (Nervous system disorders) | 7 | 1 | 8
somnolence (Nervous system disorders) | 6 | 1 | 7
facial paresis (Nervous system disorders) | 4 | 2 | 6
lymphocyte count decreased (Investigations) | 42 | 22 | 64
platelet count decreased (Investigations) | 32 | 26 | 58
white blood cell count decreased (Investigations) | 22 | 18 | 40
alanine aminotransferase increased (Investigations) | 21 | 13 | 34
aspartate aminotransferase increased (Investigations) | 18 | 8 | 26
neutrophil count decreased (Investigations) | 11 | 11 | 22
blood creatinine increased (Investigations) | 14 | 2 | 16
blood bilirubin increased (Investigations) | 10 | 2 | 12
blood alkaline phosphatase increased (Investigations) | 7 | 2 | 9
hyperglycemia (Metabolism and nutrition disorders) | 44 | 20 | 64
hypocalcaemia (Metabolism and nutrition disorders) | 36 | 14 | 50
hypoalbuminaemia (Metabolism and nutrition disorders) | 30 | 15 | 45
hypokalaemia (Metabolism and nutrition disorders) | 27 | 14 | 41
hyponatraemia (Metabolism and nutrition disorders) | 23 | 12 | 35
decreased appetite (Metabolism and nutrition disorders) | 8 | 5 | 13
hyperkalaemia (Metabolism and nutrition disorders) | 5 | 5 | 10
hypernatraemia (Metabolism and nutrition disorders) | 9 | 1 | 10
hypoglycaemia (Metabolism and nutrition disorders) | 6 | 3 | 9
fatigue (General disorders) | 53 | 14 | 67
pain (General disorders) | 26 | 7 | 33
gait disturbance (General disorders) | 11 | 2 | 13
oedema peripheral (General disorders) | 7 | 5 | 12
influenza like illness (General disorders) | 3 | 4 | 7
anaemia (Blood and lymphatic system disorders) | 48 | 20 | 68
nausea (Gastrointestinal disorders) | 19 | 8 | 27
diarrhoea (Gastrointestinal disorders) | 10 | 9 | 19
constipation (Gastrointestinal disorders) | 14 | 3 | 17
stomatitis (Gastrointestinal disorders) | 5 | 6 | 11
vomiting (Gastrointestinal disorders) | 5 | 3 | 8
gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 | 1 | 7
anal incontinence (Gastrointestinal disorders) | 3 | 3 | 6
confusional state (Psychiatric disorders) | 23 | 5 | 28
insomnia (Psychiatric disorders) | 18 | 8 | 26
agitation (Psychiatric disorders) | 8 | 3 | 11
depression (Psychiatric disorders) | 7 | 3 | 10
anxiety (Psychiatric disorders) | 7 | 2 | 9
hypertension (Vascular disorders) | 45 | 13 | 58
embolism (Vascular disorders) | 9 | 4 | 13
cough (Respiratory, thoracic and mediastinal disorders) | 10 | 1 | 11
epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 | 4 | 11
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 2 | 10
dysphonia (Respiratory, thoracic and mediastinal disorders) | 8 | 1 | 9
rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 8
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 7
oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 7
urinary tract infection (Infections and infestations) | 11 | 2 | 13
upper respiratory tract infection (Infections and infestations) | 8 | 4 | 12
muscular weakness (Musculoskeletal and connective tissue disorders) | 13 | 5 | 18
arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 3 | 8
back pain (Musculoskeletal and connective tissue disorders) | 5 | 1 | 6
urinary incontinence (Renal and urinary disorders) | 4 | 8 | 12
proteinuria (Renal and urinary disorders) | 8 | 2 | 10
haematuria (Renal and urinary disorders) | 5 | 4 | 9
pollakiuria (Renal and urinary disorders) | 7 | 1 | 8
rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 | 3 | 8
rash (Skin and subcutaneous tissue disorders) | 4 | 3 | 7
fall (Injury, poisoning and procedural complications) | 15 | 1 | 16
vision blurred (Eye disorders) | 10 | 2 | 12
sinus tachycardia (Cardiac disorders) | 8 | 5 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review. The sponsor cannot extend the embargo. The sponsor can require changes to the communication with respect to confidential information that is not necessary for the complete and accurate presentation and interpretation of the study results.

DOCUMENTS (2):
  • Study Protocol (2020-02-07): https://cdn.clinicaltrials.gov/large-docs/78/NCT02986178/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-27): https://cdn.clinicaltrials.gov/large-docs/78/NCT02986178/SAP_001.pdf